CLINICAL TRIAL: NCT01217723
Title: A Randomized Trial of Thymoglobulin to Prevent Chronic Graft Versus Host Disease in Patients Undergoing Hematopoietic Progenitor Cell Transplantation (HPCT) From Unrelated Donors
Brief Title: Thymoglobulin in Unrelated Hematopoietic Progenitor Cell Transplantation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Genzyme, a Sanofi Company (Industry); The Canadian Blood and Marrow Transplant Group (Network)
Responsible Party: Dr. Irwin Walker (Study Chair), McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CBMTG 0801
Record Dates: First submitted 2010-09-29; First posted 2010-10-08 (Estimated); Last update posted 2010-10-08 (Estimated); Status verified 2010-09

CONDITIONS: Hematologic Malignancies
Keywords: Acute leukemia (myeloid,lymphoid,or biphenotypic); Chronic myeloid leukemia; Chronic lymphocytic leukemia; Lymphoma; Myelodysplastic syndrome; Myeloproliferative disorder
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma; Myelodysplastic Syndromes; Myeloproliferative Disorders | interventions — Antilymphocyte Serum; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thymoglobulin (Experimental): Thymoglobulin will be administered on Days -2, -1 prior to the transplant and on the day of transplant.
  Interventions: Biological: Anti-Thymocyte Globulin (Rabbit)
- No Thymoglobulin (Other): Patients will receive a standard preparative regimen. (i.e. one that does not normally contain Thymoglobulin.)
  Interventions: Other: Patients will receive a standard preparative regimen (i.e. one that does not contain Thymoglobulin)

INTERVENTIONS:
Biological: Anti-Thymocyte Globulin (Rabbit) — Thymoglobulin 0.5 mg/kg on Day -2 prior to the Transplant, 2.5 mg/kg on Day -1, and 2.5 mg/kg on the day of transplant.
  Other Names: Thymoglobulin; ATGr; rabbit
  Arms: Thymoglobulin
Other: Patients will receive a standard preparative regimen (i.e. one that does not contain Thymoglobulin) — The standard preparative regimen can be myeloablative or reduced intensity.
  Arms: No Thymoglobulin

SUMMARY:
This is a randomized trial for patients undergoing hematopoietic progenitor cell transplantation (HPCT) from an unrelated donor. Approximately 50% of the patients enrolled will receive Thymoglobulin® as part of the preparative regimen prior to HPCT. The other 50% of the patients enrolled will receive a standard preparative regimen. Thymoglobulin is known to suppress the types of cells that can cause a transplant complication known as "chronic graft versus host disease (cGVHD)". The goal of this trial is to find out if adding Thymoglobulin to the preparative regimen will result in a decrease in cGVHD.

DETAILED DESCRIPTION:
This study is a non-blinded, randomized, multicentre trial testing the effect of Thymoglobulin® vs. placebo on the primary outcome of cGVHD. Subjects will be children and adults having unrelated donor transplants.

Intervention: Infusion of Thymoglobulin® on three days prior to the transplant.

Hypothesis: The hypothesis is that the use of Thymoglobulin® in the experimental group will result in an absolute 20% increase in the number of patients free of cGVHD at 12 months, the time of peak incidence, from 20% in the control group to 40% in the experimental group.

Outcome Measures: The Primary Outcome Measure is freedom from cGVHD at 12 months from transplantation, defined as withdrawal of all systemic immunosuppressive agents and without resumption up to 12 months (a binary end-point, yes/no). Secondary outcome measures: Quality of Life, overall incidence of cGVHD (including untreated cases and resolved cases), the incidence of "extensive" cGVHD, time to non-relapse mortality, time to all-cause mortality, time to relapse of leukemia, graft rejection or failure (Yes vs. No), serious infection (Yes vs. No), CMV activation (Yes vs. No), organ-specific grading of chronic graft versus host disease, resumption of immunosuppressive agents after 12 months (Yes vs. No), doses of immunosuppressive drugs still required at 12 months, and incidence of acute graft versus host disease.

ELIGIBILITY:
Inclusion Criteria:

* The recipient has a hematologic malignancy
* The recipient will receive one of the specified preparative regimens
* The recipient will receive either a bone marrow ("HPC, Marrow") or blood progenitor cell ("HPC, Apheresis") graft
* The recipient has an unrelated donor who with high resolution typing is either fully MHC matched at HLA-A, B, C and DRB1 with the recipient or is 1-antigen or 1-allele mismatched at A, B, C or DRB1 loci The recipient meets the transplant centre's criteria for unrelated donor allogeneic transplantation , either myeloablative or non-myeloablative (syn. RIC).
* The recipient has good performance status (Karnofsky ≥60%)
* Recipient has given signed informed consent For the questionnaire component only, be able to complete the questionnaires in English or with a validated translation (as posted on the project website)

Exclusion Criteria:

* The recipient is HIV antibody positive
* The recipient has a hypersensitivity to rabbit proteins or Thymoglobulin pharmaceutical excipients, glycine or mannitol
* The recipient has active or chronic infection (i.e. infection requiring oral or IV therapy)
* The recipient (if female and of childbearing potential) is pregnant or breast-feeding at the time of enrollment
* The recipient (if female and of childbearing potential) does not agree to use an adequate contraceptive method from the time of enrollment until a minimum of one year following transplant
* The recipient (if male and fertile) does not agree to use an adequate contraceptive method from the time of enrollment until a minimum of one year following transplant
* For the questionnaire component only, the recipient is unable to participate due to cognitive, linguistic or emotional difficulties (i.e. the recipient can participate in the main study but will be excluded from the questionnaire component

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2010-04; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from Chronic GVHD | 12 months post transplant
  "Freedom from Chronic GVHD" is defined as withdrawal of all systemic immunosuppressive agents and without resumption up to 12 months (a binary endpoint, yes/no)

SECONDARY OUTCOMES:
Quality of Life | Measured at Screening, Month 6, 12 and 24
  A series of questionnaires measured at the screening interval (up to 3 months prior to transplant), 6, 12 and 24 months post transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Irwin Walker, MD, Study Chair — McMaster University, Faculty of Health Sciences
Locations (10):
- Canada (10):
  - Vancouver General Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Juravinski Hospital & Cancer Centre, Hamilton, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital de l'Enfant Jesus, Montreal, Quebec
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
  - L'Hotel Dieu de Quebec, Québec, Quebec

REFERENCES:
- [Derived] Chakupurakal G, Freudenberger P, Skoetz N, Ahr H, Theurich S. Polyclonal anti-thymocyte globulins for the prophylaxis of graft-versus-host disease after allogeneic stem cell or bone marrow transplantation in adults. Cochrane Database Syst Rev. 2023 Jun 21;6(6):CD009159. doi: 10.1002/14651858.CD009159.pub3. PMID 37341189
- [Derived] Walker I, Panzarella T, Couban S, Couture F, Devins G, Elemary M, Gallagher G, Kerr H, Kuruvilla J, Lee SJ, Moore J, Nevill T, Popradi G, Roy J, Schultz KR, Szwajcer D, Toze C, Foley R; Cell Therapy Transplant Canada. Addition of anti-thymocyte globulin to standard graft-versus-host disease prophylaxis versus standard treatment alone in patients with haematological malignancies undergoing transplantation from unrelated donors: final analysis of a randomised, open-label, multicentre, phase 3 trial. Lancet Haematol. 2020 Feb;7(2):e100-e111. doi: 10.1016/S2352-3026(19)30220-0. Epub 2020 Jan 17. PMID 31958417
- [Derived] Naeije L, Kariminia A, Abdossamadi S, Azadpour S, Subrt P, Kuzeljevic B, Irvine MA, Walker I, Schultz KR. Anti-Thymocyte Globulin Prophylaxis Induces a Decrease in Naive Th Cells to Inhibit the Onset of Chronic Graft-versus-Host Disease: Results from the Canadian Bone Marrow Transplant Group (CBMTG) 0801 Study. Biol Blood Marrow Transplant. 2020 Mar;26(3):438-444. doi: 10.1016/j.bbmt.2019.11.015. Epub 2019 Nov 19. PMID 31756535